CLINICAL TRIAL: NCT05697445
Title: Combined Effect Of Cranial And Cervical Mobilization In Patients With Cervicogenic Headache
Brief Title: Combined Effect Of Cranial And Cervical Mobilization In Patients With CGH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennat Allah Hussien Mahmoud Mouhamed, physical therapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mobilization In CGH Treatment
Record Dates: First submitted 2022-12-29; First posted 2023-01-25 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Cervicogenic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cranial Mobilization and Exercises Group (Experimental)
  Interventions: Other: Mobilization Techniques; Other: Conventional Treatment
- Exercises Group (Active Comparator)
  Interventions: Other: Conventional Treatment

INTERVENTIONS:
Other: Mobilization Techniques — Combination of Cranial and Cervical Mobilization for Cervicogenic headache Patients treatment
  Arms: Cranial Mobilization and Exercises Group
Other: Conventional Treatment — Cervicogenic headache exercises

SUMMARY:
* The purposes of this study are:
* To investigate the combined effect of cranial and cervical mobilization in patient with cervicogenic headache and there effect on :

  1. Perceptive neck pain intensity
  2. Perceptive headache intensity
  3. pain by pressure
  4. frequency of headache episodes
  5. duration of headache episodes
  6. Medications uptakes

ELIGIBILITY:
Inclusion Criteria:

* pain originating at the neck and radiating to oculo-frontal-temporal regions.
* symptom unilaterally.
* symptom provocation through cervical movement and/or awkward cervical postural.
* symptom provocation through external pressure application through palpation to associated posterior cervical spine segments with resultant symptom reproduction.
* possible ipsilateral shoulder and/or arm pain of vague reference.
* 15 or more headache episodes per month
* No history of cervical operation or any disease that result in headache as colities -All patients will sign the informed consent before joining the study.

Exclusion Criteria:

* Headache not of cervical origin
* Headache with autonomic involvement, dizziness, or visual disturbance
* Congenital conditions of the cervical spine
* It is of primary concern to exclude serious or life-threatening pathology such as :
* cranial tumors.
* Meningitis.
* sub-arachnoid hemorrhage.
* carotid artery,vertebral artery dissection.
* History of cervical operation or any disease that result in headache as colitis
* Age less than 18 or more than 40 years
* chronic maxillary sinusitis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Assis Headache Perceptive intensity | 2 weeks
  By visual analog scale , Minimum value zero mean No pain Maximum value 10 mean Worst pain .